CLINICAL TRIAL: NCT06826274
Title: Clinical and Neurophysiological Evaluation of the Effects of Cervical TsDCS on Stroke Patients with Distal Upper Limb Strength Deficit
Brief Title: Cervical TsDCS on Stroke Patients
Acronym: AMPLI-MOV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RP 23/06
Record Dates: First submitted 2025-01-29; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Functional Recovery; Motor Rehabilitation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stroke (Experimental)
  Interventions: Other: tDCS
- Healthy (Experimental)
  Interventions: Other: tDCS

INTERVENTIONS:
Other: tDCS — Transcranial direct current stimulation

SUMMARY:
The present project aims to evaluate the facilitatory modulation of motor responses of the limb upper limb by tsDCS in patients with arm/hand hyposthenia after cerebral ischemia to verify the possible therapeutic benefits that this type of stimulation can induce in terms of of strength, dexterity and effectiveness in acts of daily living.

ELIGIBILITY:
Group Stroke:

Inclusion criteria:

1. age over 18 years;
2. first ischemic/hemorrhagic stroke (within 30 days of onset);
3. mild-to-moderate stroke (NIHSS scale score<16).
4. residual function of the upper limb, assessed by the following scales: - MRC of the distal muscles of the upper limb: score between 2 and 4; - NHISS (items 5A and 5B): score between 1 and 3;
5. ability to give informed consent and understand instructions.

Exclusion criteria:

1. severe spasticity (Ashworth Scale score > 2);
2. severe aphasia;
3. severe neglect;
4. history of disabling neurological disease;
5. history of epilepsy;
6. significant comorbidities;
7. contraindications to tsDCS.

Healthy Group:

Inclusion criteria:

1. age over 18 years;
2. equalized in age with the patient group.

Exclusion criteria:

1. history of stroke progress;
2. history of severe neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
improvement of paretic hand performance | through study completion, an average of 1 year
  The primary outcome measure is the improvement in hand strength and dexterity in individuals with upper limb motor impairment following cerebral ischemia, after the application of tsDCS at the cervical spinal level during Reaching
improvement of paretic hand performance | through study completion, an average of 1 year
  The primary outcome measure is the improvement in hand strength and dexterity in individuals with upper limb motor impairment following cerebral ischemia, after the application of tsDCS at the cervical spinal level during Grasping
improvement of paretic hand performance | through study completion, an average of 1 year
  The primary outcome measure is the improvement in hand strength and dexterity in individuals with upper limb motor impairment following cerebral ischemia, after the application of tsDCS at the cervical spinal level during Lifting test
improvement of paretic hand performance | through study completion, an average of 1 year
  The primary outcome measure is the improvement in hand strength and dexterity in individuals with upper limb motor impairment following cerebral ischemia, after the application of tsDCS at the cervical spinal level duringthe Nine Hole Peg test
improvement of paretic hand performance | through study completion, an average of 1 year
  The primary outcome measure is the improvement in hand strength and dexterity in individuals with upper limb motor impairment following cerebral ischemia, after the application of tsDCS at the cervical spinal level during finger mobility tests

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Roma, Rome, Rome, Italy